CLINICAL TRIAL: NCT01483950
Title: Non-interventional Study to Assess Reaching of Cholesterol Target Values in Patients Treated With HMG-CoA Reductase Inhibitors in Bosnia and Herzegovina
Brief Title: Evaluation of Patients Treated With HMG-CoA Reductase Inhibitors to Reach Cholesterol Target Values
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CBA-CRE-2011/1
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Hypercholesterolaemia
Keywords: Dyslipidemia; Statins; Total Cholesterol; Low density lipoprotein (LDL) cholesterol; High density lipoprotein (HDL) cholesterol
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with hypercholesterolaemia

SUMMARY:
This study is non-interventional study of patients who are treated with any HMGCoA reductase inhibitors (rosuvastatin, simvastatin,atorvastatin and fluvastatin) available in Bosnia and Herzegovina for at least 6 months. Data collection for each patient will take place at a single visit. The investigators will complete Case Report Form (CRF) with patient's demographic, the presence of the factors for high cardiovascular risk, current treatment, cholesterol value as well as with further treatment decision.

DETAILED DESCRIPTION:
Non-interventional study to assess reaching of cholesterol target values in patients treated with HMG-CoA reductase inhibitors in Bosnia and Herzegovina

ELIGIBILITY:
Inclusion Criteria:

* Patients, treated with one HMG-CoA reductase inhibitors for at least 6 months without changing the dose for the last 4 weeks at least
* All patients must sign informed consent form

Exclusion Criteria:

* Patients who have not signed the Informed Consent Form
* Patients with contraindication for the treatment with HMG-CoA reductase inhibitors as per SmPC approved in Bosnia and Herzegovina

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated by specialist
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The number and percentage of patients reaching the LDL-C goals, according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated

SECONDARY OUTCOMES:
The number and percentage of patients reaching the total cholesterol goals, according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
The number and percentage of patients with high cardiovascular risk reaching the LDL-C goals, according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated
The number and percentage of patients with high cardiovascular risk reaching the total cholesterol goals, according to the Fourth Joint European Task Force guideline. | During the study visit scheduled at least 6 months after HMG-CoA reductase inhibitor has been initiated

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Loza, DOC. DR. SCI. MED, Principal Investigator — Klinika za bolesti srca i reumatizma Sarajevo , Bosnia and Herzegovina; Meta Jeras, MR PH, Study Director — West Balkan MD
Locations (14):
- Bosnia and Herzegovina (14):
  - Research Site, Banja Luka
  - Research Site, Bijeljina
  - Research Site, Doboj
  - Reserach Site, Gradiška
  - Research Site, Kakanj
  - Research Site, Maglaj
  - Research Site, Prijedor
  - Research Site, Sarajevo
  - Research Site, Tešanj
  - Research Site, Trebinje
  - Research Site, Visoko
  - Research Site, Zavidovići
  - Research Site, Zenica
  - Research Site, Zvornik